CLINICAL TRIAL: NCT05921006
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food-effect of Single and Multiple Oral Doses of RJ4287 in Healthy Volunteers
Brief Title: Ascending Single-Dose and Multiple-Dose Study to Evaluate RJ4287 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Ruijie Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RJ4287001
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Drug Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RJ4287 Tablets (Experimental): single-dose or Multiple-doses, ascending dosing groups (cohorts) will be evaluated
  Interventions: Drug: RJ4287
- Placebo (Placebo Comparator): Single or multiple doses of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RJ4287 — Oral，tablets，Once daily for 14 days
  Arms: RJ4287 Tablets
Drug: Placebo — Oral，tablets，Once daily daily for 14 days
  Arms: Placebo

SUMMARY:
A Randomized Study of RJ4287 Drug to Evaluate the Safety, Tolerability, Pharmacokinetics and Food-effect of Single and Multiple Doses in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male and Female between 18 and 55 years old，inclusive
* Body weight >50 kg for Male and >45 kg for Female with a body mass index BMI between 19-28 kg/m2（inclusive）
* Female subjects of childbearing potential who have had no unprotected sex within 14 days prior to screening and who have had a negative pregnancy test during the screening period; subjects (including partners) who have no plans for pregnancy, sperm donation or egg donation and are willing to use effective contraception from the time of informed consent until 6 months after administration of the test product;
* The subject must be willing and able to provide written informed consent

Exclusion Criteria:

* History of thyroid disorder or abnormal thyroid function tests at screening
* Abnormal abdominal ultrasound findings with clinical significance
* Subjects with any of the following laboratory tests at screening or baseline were not eligible for enrollment in this study: 1) Glutamic transaminase (AST), glutamic aminotransferase (ALT) or direct bilirubin above the upper limit of the reference range at screening; 2) Positive screening for HIV antibodies, hepatitis B surface antigen, hepatitis C antibodies, syphilis antibodies ECG QTc > 450 ms, QRS > 110 ms, intermittent bundle branch block, frequent premature atrial or ventricular contractions at the time of screening, or any person who is considered clinically significant by the investigator; 4) A routine blood test with a white blood cell count, neutrophil count and lymphocyte count outside the normal reference range at screening and judged clinically significant by the investigator; 5) A kidney disease diet adjustment ( MDRD) formula calculated with an estimated glomerular filtration rate (eGFR) < 90 mL
* Sensitivity to thyroid medication or history of sensitivity to a similar study drug(eg.MGL-3196)
* History of sensitivity to a similar study drug
* Major surgical procedure, previous gastrointestinal surgery, vagotomy, bowel resection or any surgical procedure that may interfere with peristalsis, pH or absorption in the gastrointestinal tract within 6 months prior to screening
* Subjects who, in the judgement of the investigator, have a condition that affects the absorption, distribution, metabolism and excretion of the drug (e.g. gastrointestinal dysfunction, peptic ulcer, gastrointestinal surgery, etc.) or who are unable to comply with a uniform diet during the trial
* Taken any prescription medication, over-the-counter medication, any vitamin product or herbal remedy within 1 month prior to screening
* Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results interpretation
* History of regular use nicotine or alcohol，unable to abstain from smoking and alcohol during the trial
* Previous blood donation or blood loss of more than 400 mL within 3 months prior to taking the study drug
* Had consumed a special diet (including popcorn, dragon fruit, mango, grapefruit, orange, etc.) or alcohol within 2 weeks before taking the study drug, or had strenuous exercise
* Taken an experimental drug or other experimental treatment within 3 months prior to screening, or being involved in any other interventional clinical trial
* Nursing female subjects
* Any other condition that, in the opinion of the investigator or sponsor, makes the subject unsuitable for inclusion in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 month
  Safety measurements will include vital signs, hematology, blood chemistry, blood pressure and other readouts.

SECONDARY OUTCOMES:
Pharmacokinetics parameters of blood | 2 weeks
  To measure the plasma concentration of RJ4287 in single and multiple doses
Pharmacokinetics parameters of urine | 2 weeks
  Accumulated excretion
Pharmacokinetics parameters of faeces | 2 weeks
  Accumulated excretion
Change in lipid / lipoprotein levels from baseline through Day 14 in Multiple Dose | 2 weeks
  compare with placebo

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alkhouri N. Thyromimetics as emerging therapeutic agents for nonalcoholic steatohepatitis: rationale for the development of resmetirom (MGL-3196). Expert Opin Investig Drugs. 2020 Feb;29(2):99-101. doi: 10.1080/13543784.2020.1708899. Epub 2019 Dec 25. No abstract available. PMID 31868036
- [Background] Taub R, Chiang E, Chabot-Blanchet M, Kelly MJ, Reeves RA, Guertin MC, Tardif JC. Lipid lowering in healthy volunteers treated with multiple doses of MGL-3196, a liver-targeted thyroid hormone receptor-beta agonist. Atherosclerosis. 2013 Oct;230(2):373-80. doi: 10.1016/j.atherosclerosis.2013.07.056. Epub 2013 Aug 21. PMID 24075770
- [Background] Harrison SA, Bashir MR, Guy CD, Zhou R, Moylan CA, Frias JP, Alkhouri N, Bansal MB, Baum S, Neuschwander-Tetri BA, Taub R, Moussa SE. Resmetirom (MGL-3196) for the treatment of non-alcoholic steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2019 Nov 30;394(10213):2012-2024. doi: 10.1016/S0140-6736(19)32517-6. Epub 2019 Nov 11. PMID 31727409